CLINICAL TRIAL: NCT02709759
Title: Behavioral Interventions to Reduce Heavy Drinking Among MSM in HIV Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Christopher W. Kahler, Professor, Brown University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: P01AA01907
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Results first posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-04

CONDITIONS: Alcohol Drinking; HIV
MeSH Terms: conditions — Alcohol Drinking | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- MI (Active Comparator): Motivational interviewing focused on reducing alcohol use, delivered by videoconferencing.
  Interventions: Behavioral: Motivational intervention
- BA (Active Comparator): Brief Advice to reduce drinking delivered by videoconferencing
  Interventions: Behavioral: Brief Advice
- MI + ITM (Active Comparator): Motivational intervention to reduce drinking, delivered by videoconferencing, plus Interactive text messaging around alcohol use
  Interventions: Behavioral: Motivational intervention; Behavioral: Interactive text messaging
- BA + ITM (Active Comparator): Brief Advice to reduce drinking, delivered by videoconferencing, plus Interactive text messaging around alcohol use
  Interventions: Behavioral: Brief Advice; Behavioral: Interactive text messaging
- MI + ITM + EI (Active Comparator): Participants in this arm receive MI delivered by videoconferencing and ITM over 9 months rather than 1
  Interventions: Behavioral: Motivational intervention; Behavioral: Interactive text messaging
- BA + ITM + EI (Active Comparator): Participants in this arm receive BA delivered by videoconferencing and ITM over 9 months rather than 1
  Interventions: Behavioral: Brief Advice; Behavioral: Interactive text messaging
- BA + EI (Active Comparator): Participants in this arm receive BA delivered by videoconferencing over 9 months rather than 1
  Interventions: Behavioral: Brief Advice; Behavioral: Interactive text messaging
- MI + EI (Active Comparator): Participants in this arm receive MI delivered by videoconferencing over 9 months rather than 1
  Interventions: Behavioral: Motivational intervention; Behavioral: Interactive text messaging

INTERVENTIONS:
Behavioral: Motivational intervention — Involves 60 minutes of counseling delivered by videoconferencing. Provides feedback on drinking and HIV and related behaviors.
  Arms: MI; MI + EI; MI + ITM; MI + ITM + EI
Behavioral: Brief Advice — Involves 5-10 minutes of brief counseling to reduce drinking
  Arms: BA; BA + EI; BA + ITM; BA + ITM + EI
Behavioral: Interactive text messaging — Involves receiving daily text messages that enable participants to track their drinking and related consequences. Provides feedback on drinking and allow setting of goals.
  Arms: BA + EI; BA + ITM; BA + ITM + EI; MI + EI; MI + ITM; MI + ITM + EI

SUMMARY:
The purpose of the present study is to conduct a fully-crossed 2 X 2 X 2 factorial randomized controlled trial with a diverse sample of 224 MSM recruited from 2 urban HIV primary care clinics (one in the Northeast and one in the South). The first study factor will compare brief advice (BA) vs. a motivational intervention (MI) that contains detailed personalized normative and HIV-specific feedback. The second factor compares an interactive text messaging (ITM) intervention vs. no text messaging. The final factor compares intervention of low intensity and duration (two sessions over 1 month) to extended intervention (EI) entailing 5 sessions over 9 months.

DETAILED DESCRIPTION:
Heavy drinking in HIV-infected patients can lead to low antiretroviral therapy adherence and poor virologic control, greater sexual risk taking, increased risk of liver disease, and decreased cognitive function. Therefore, reductions in drinking may have particularly positive and widespread effects in HIV-infected patients. Men who have sex with men (MSM) continue to represent the majority of new HIV infections, and HIV-infected MSM have rates of hazardous drinking as high as 33%. Therefore, developing and testing interventions to reduce heavy drinking in HIV-infected MSM is a very high public health priority. There have been relatively few alcohol interventions tested that focus on MSM, and only two have addressed drinking in HIV-infected MSM. Although recent studies indicate that behavioral interventions can reduce heavy drinking in HIV-infected patients, much remains unknown about the efficacy of different approaches to behavioral intervention and their unique and combined effects. The purpose of the present study is to conduct a fully-crossed 2 X 2 X 2 factorial randomized controlled trial with a diverse sample of 224 MSM recruited from 2 urban HIV primary care clinics (one in the Northeast and one in the South). The first study factor will compare brief advice (BA) vs. a motivational intervention (MI) that contains detailed personalized normative and HIV-specific feedback. The second factor compares an interactive text messaging (ITM) intervention vs. no text messaging. The final factor compares intervention of low intensity and duration (two sessions over 1 month) to extended intervention (EI) entailing 5 sessions over 9 months. BA and MI will be delivered by a core set of interventionists from a central location using a webcam-enabled telemedicine system, which can facilitate larger-scale implementation. The design will allow us to test the hypothesis that MI compared to BA, ITM compared to no ITM, and EI compared to no EI, will result in significantly greater reductions in number of alcoholic drinks consumed and number of heavy drinking days at 6- and 12-month follow-ups. Secondary outcomes include engagement in unprotected anal intercourse, ART adherence and viral suppression, CD4 cell count, liver function tests, and neurocognitive function. We also will test the hypothesis that the effects of MI, ITM, and EI on drinking will be moderated by alcohol use disorder status and readiness to change drinking such that these interventions will be relatively more efficacious in those with a current disorder and those with low readiness. The study will provide crucial evidence regarding which intervention approaches, alone or in combination, are likely to be most efficient to implement on a large scale in HIV care settings.

ELIGIBILITY:
Inclusion Criteria:

* be at least 18 years of age
* drink heavily at least once per month on average (≥5 drinks) or drink have drunk more than 14 drinks per week over the past 3 months
* have a confirmed diagnosis of HIV
* be a biological male who identifies as male
* report having had sex (oral or anal) with a male partner in the past 12 months and/or, identify as gay or bisexual.
* For those on ART, they must be stabilized on their current regimen for at least 3 months prior to study enrollment.

Exclusion Criteria:

* report past 3 month intravenous drug use
* are currently psychotic, suicidal, or manic
* being treated or have been treated in the past 3 months for an HIV-related opportunistic infection
* currently receiving treatment for an alcohol or drug problem.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2022-01-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Fenway Health, Boston, Massachusetts
  - Center for Alcohol and Addiction Studies, Brown University, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kahler CW, Surace A, Liu T, Pantalone DW, Mastroleo NR, Yan Y, Wray TB, Mayer KH, Monti PM. Efficacy of Behavioral Intervention, Text Messaging, and Extended Intervention to Address Alcohol Misuse in Sexual Minority Men with HIV: A Factorial Randomized Clinical Trial. AIDS Behav. 2024 Dec;28(12):3970-3983. doi: 10.1007/s10461-024-04493-x. Epub 2024 Sep 13. PMID 39266891

RESULTS

PARTICIPANT FLOW:
Groups:
- MI Only: Motivational interviewing focused on reducing alcohol use, delivered by videoconferencing.
  Motivational intervention: Involves 60 minutes of counseling delivered by videoconferencing. Provides feedback on drinking and HIV and related behaviors.
- BA Only: Brief Advice to reduce drinking delivered by videoconferencing
  Brief Advice: Involves 5-10 minutes of brief counseling to reduce drinking
Period: Overall Study
Arm/Group | MI Only | BA Only | MI + ITM | BA + ITM | MI + ITM + EI | BA + ITM + EI | BA + EI | MI + EI
Started | 24 | 24 | 23 | 23 | 23 | 23 | 24 | 24
Completed | 16 | 16 | 18 | 18 | 14 | 16 | 16 | 16
Not Completed | 8 | 8 | 5 | 5 | 9 | 7 | 8 | 8

BASELINE CHARACTERISTICS:
Groups:
- Motivational Interviewing (MI): Motivational interviewing focused on reducing alcohol use, delivered by videoconferencing.
  Motivational intervention: Involves 60 minutes of counseling delivered by videoconferencing. Provides feedback on drinking and HIV and related behaviors.
- Brief Advice (BA): Brief Advice to reduce drinking delivered by videoconferencing
  Brief Advice: Involves 5-10 minutes of brief counseling to reduce drinking
- Total: Total of all reporting groups
Arm/Group | Motivational Interviewing (MI) | Brief Advice (BA) | MI + ITM | BA + ITM | MI + ITM + EI | BA + ITM + EI | BA + EI | MI + EI | Total
Number analyzed (Participants) | 24 | 24 | 23 | 23 | 23 | 23 | 24 | 24 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (9.4) | 47.8 (8.1) | 46.7 (11.9) | 48.0 (13.4) | 51.2 (9.3) | 21.7 (9.8) | 49.3 (12.2) | 51.0 (9.5) | 49.3 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 24 | 24 | 23 | 23 | 23 | 23 | 24 | 24 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 6 | 4 | 9 | 4 | 6 | 4 | 8 | 47
  Not Hispanic or Latino | 18 | 18 | 19 | 14 | 19 | 17 | 20 | 16 | 141
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 16 | 13 | 15 | 12 | 14 | 18 | 12 | 12 | 112
  White | 7 | 9 | 6 | 9 | 7 | 5 | 10 | 11 | 64
  More than one race | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2
Alcoholic drinks per week [Mean (Standard Deviation); unit: Alcohol drinks] | 27.1 (19.2) | 23.4 (18.2) | 24.3 (16.9) | 19.1 (19.8) | 20.7 (14.7) | 28.6 (26.2) | 26.3 (21.4) | 35.7 (35.8) | 25.7 (22.6)
Number of heavy drinking days [Mean (Standard Deviation); unit: days] — Days drinking 5 or more drinks in the past 30 days
  days | 11.8 (10.2) | 8.4 (8.9) | 10.5 (10.0) | 7.4 (8.7) | 8.8 (7.5) | 10.5 (10.1) | 12.0 (11.8) | 10.7 (10.1) | 10.0 (9.7)

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Drinks Per Week at 6 Months
Description: Average number of alcoholic drinks consumed per week assessed at 6 months. Covers the period of 30 days prior to the assessment.
Time Frame: Past 30 days
Measure: Mean (Standard Deviation); unit: number of drinks
Arm/Group | Motivational Interviewing (MI) | Brief Advice (BA) | MI + ITM | BA + ITM | MI + ITM + EI | BA + ITM + EI | BA + EI | MI + EI
Number analyzed (Participants) | 23 | 17 | 19 | 22 | 17 | 16 | 14 | 19
number of drinks | 13.3 (14.7) | 14.9 (17.4) | 7.5 (8.7) | 5.0 (5.9) | 9.6 (10.2) | 7.6 (12.2) | 7.7 (9.3) | 17.8 (22.5)

2. Primary Outcome: Average Number of Alcoholic Drinks Consumed Per Week Assessed at 12 Months
Description: Average number of alcoholic drinks consumed per week assessed at 12 months. Covers the period of 30 days prior to the assessment.
Time Frame: Past 30 days
Measure: Mean (Standard Deviation); unit: number of drinks
Arm/Group | Motivational Interviewing (MI) | Brief Advice (BA) | MI + ITM | BA + ITM | MI + ITM + EI | BA + ITM + EI | BA + EI | MI + EI
Number analyzed (Participants) | 16 | 16 | 18 | 18 | 14 | 16 | 17 | 18
number of drinks | 8.3 (7.2) | 16.5 (17.0) | 4.6 (5.9) | 3.7 (5.3) | 5.4 (7.1) | 8.1 (9.9) | 7.0 (8.9) | 11.6 (13.4)

3. Primary Outcome: Number of Heavy Drinking Days at 6 Months
Description: Number of heavy drinking days (5 or more alcoholic drinks in a single day) assessed at 6 months
Time Frame: Past 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MI Only | BA Only | MI + ITM | BA + ITM | MI + ITM + EI | BA + ITM + EI | BA + EI | MI + EI
Number analyzed (Participants) | 23 | 17 | 19 | 22 | 17 | 16 | 14 | 19
Days | 4.3 (5.8) | 5.2 (8.1) | 1.8 (2.7) | 1.4 (2.3) | 3.1 (5.0) | 3.5 (7.7) | 1.6 (3.4) | 6.1 (9.9)

4. Primary Outcome: Number of Heavy Drinking Days at 12 Months
Description: Number of days drinking 5 or more alcoholic drinks
Time Frame: Past 30 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Motivational Interviewing (MI) | Brief Advice (BA) | MI + ITM | BA + ITM | MI + ITM + EI | BA + ITM + EI | BA + EI | MI + EI
Number analyzed (Participants) | 16 | 16 | 18 | 18 | 14 | 16 | 17 | 18
Days | 2.2 (2.7) | 5.6 (9.6) | 1.8 (3.4) | 1.2 (3.0) | 2.6 (4.9) | 2.7 (4.0) | 2.4 (4.5) | 3.8 (6.7)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | MI Only | BA Only | MI + ITM | BA + ITM | MI + ITM + EI | BA + ITM + EI | BA + EI | MI + EI
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/23 | 0/23 | 0/23 | 0/23 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/23 | 0/23 | 0/23 | 0/23 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/23 | 0/23 | 0/23 | 0/23 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/59/NCT02709759/Prot_SAP_000.pdf